CLINICAL TRIAL: NCT00805714
Title: A Prospective Clinical Observation Study to Evaluate the Influence of Long Term Treatment of Pitavastatin on the Therapeutic Prognosis and Safety in Acute Myocardial Infarction
Brief Title: Livalo Acute Myocardial Infarction Study
Acronym: LAMIS
Status: Completed | Type: Observational
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: PTV-KAMI
Record Dates: First submitted 2008-12-02; First posted 2008-12-10 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute myocardial infarction: AMI patients who are in need to be treated by statins

SUMMARY:
Statins are usually used in AMI patients due to its strong anti-lipidemic effect, pleiotropic effect and tolerable safety profiles. Generally AMI patients are prescribed many drugs concomitantly; there are some risks due to the drug interaction. Especially, statins are reported to have many drug interactions, these might influence to therapeutic prognosis and safety in AMI patients.

This study is conducted to administer the non-CYP3A4 metabolized statin, pitavastatin to AMI patients over 1 year, and the results will be compared with the other results from the KAMIR study which is expected to the large scale of AMI patients using statins be enrolled. Finally, from that comparison, we will investigate the influence of the statins metabolism by CYP3A4 to the therapeutic prognosis like death, major adverse cardiac events(MACE), and major ADR of statins like CK increase, myalgia.

ELIGIBILITY:
Inclusion Criteria:

* The patients who have taken pitavastatin since AMI

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AMI patients who are in need to be treated by statins
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Death/MACE for 1 year after the registration | 1 year

SECONDARY OUTCOMES:
Achievement of LDL cholesterol target level according to the NCEP ATP III guideline | 1 year
Abnormal change of lab value including CK etc | 1 year
Adverse event including myalgia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Myung Ho Jeong, Principal Investigator — Chonnam National University Hospital
Locations (10):
- South Korea (10):
  - Cardiac and Vascular Center, Hanseo Hospital, Busan
  - Departments of Cardiology, Catholic University of Daegu College of Medicine, Daegu
  - Division of Cardiology, Department of Internal Medicine, School of Medicine, Keimyung University, Daegu
  - Division of Cardiology, Heart Center, Konyang University, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Department of Cardiovascular Medicine, Wonkwang University School of Medicine, Iksan
  - Gachon University Gil Medical Center, Incheon
  - Division of Cardiology Cardiac Center, Seoul National University Bundang Hospital, Seongnam
  - Cardiovascular Center, Korea University Guro Hospital, Seoul
  - Heart Center, Division of Cardiology, Chung-Ang University Hospital, Seoul